CLINICAL TRIAL: NCT04595643
Title: Outpatient Swallowing Therapy for Subjects With Neurological Illness - a Feasability Study
Brief Title: Outpatient Swallowing Therapy for Subjects With Neurological Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-182-20
Record Dates: First submitted 2020-09-18; First posted 2020-10-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-09

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specialized dysphagia treatment (Experimental): Dysphagia treatment is provided by occupational therapists specialized in dysphagia.
  Interventions: Other: Combination of different dysphagia training modalities

INTERVENTIONS:
Other: Combination of different dysphagia training modalities — Neuromuscular electrical stimulation, Masako exercises, Mendelsohn maneuver, chin down, mobilization, shaker exercises, eating different food consistencies.

SUMMARY:
Health care staff in the municipalities do not always have the necessary competencies to treat patients with dysphagia. At the present neurorehabilitation hospital dysphagia examinations for outpatients are provided.

The objective is to investigate the effect of a specialized outpatient dysphagia unit for subjects with dysphagia following neurological illness. Occupational therapists from the outpatient dysphagia unit will train with subjects for 2-3 weeks, and supervise furter training provided by health care staff in the municipalities.

ELIGIBILITY:
Inclusion Criteria:

* Neurological illness
* Living in the Region of central Jutland
* FEDSS score 2-6

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS) | Baseline and 14 days follow-up
  The FEDSS assess severity of dysphagia, with scores ranging 1-6. Higher scores mean worse outcome.
Change in Functional Oral Intake Scale (FOIS) | Baseline, immediately after the intervention, and 14 days follow-up
  Level of oral intake with scores ranging 1-7. Higher scores mean better outcome.

SECONDARY OUTCOMES:
Change in Penetration Aspiration Scale (PAS) | Baseline and 14 days follow-up
  Assessment of aspiration with scores ranging 1-8. Higher scores mean worse outcome.
Change in The Yale Pharyngeal Residue Severity Rating Scale | Baseline and 14 days follow-up
  Assessment of residue location and amount of residue. Two subscales with scores ranging 1-5. Higher scores mean worse outcome.
Facio Oral Tract Therapy - Swallowing assessment of Saliva (FOTT-SAS) | Baseline, immediately after the intervention, and 14 days follow-up
  Clinical examination of swallowing function. Yes or no to initiation of oral intake (binary outcome).
Dysphagia Handicap Index (DHI) | Baseline, immediately after the intervention, and 14 days follow-up
  Questionnaire on experience of dysphagia. 25 items with a toal score ranging 0-100. Higher scores mean worse outcome. Also measures overall severity with scores ranging 1-7. Higher scores means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Fabricius, PhD, Principal Investigator — Hammel Neurorehabilitation Centre and Univeristy Research Clinic
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Region of Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No